

A Prospective, Randomized, Controlled, Multi-Center Evaluation of a Powered Vascular Stapler in Laparoscopic Nephrectomies and Nephroureterectomies

Protocol #: ESC-15-002

Document Effective Date

Original November 17, 2015

**Sponsor:** 

Ethicon Endo-Surgery, Inc. 4545 Creek Road Cincinnati, OH 45242

#### **CONFIDENTIALITY STATEMENT**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. Subject to the foregoing, this information may be disclosed only to those persons involved in the study who have a need to know, but all such persons must be instructed not to further disseminate this information to others. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

Protocol ESC-15-002 



A Prospective, Randomized, Controlled, Multi-Center Evaluation of a Powered Vascular Stapler in Laparoscopic Nephrectomies and Nephroureterectomies

Protocol Number: ESC-15-002

Approval:



#### COMPLIANCE STATEMENT

This study will be conducted in compliance with Good Clinical Practice (and in accordance with the Declaration of Helsinki) as well as all applicable local regulations.



#### **INVESTIGATOR SIGNATURE**

I have read, understood, and agree to:

- Ensure that the requirements for obtaining informed consent are met;
- Conduct the study in accordance with this protocol, including applicable local laws and regulations;
- Maintain the confidentiality of all information received or developed in connection with this protocol;
- Report all serious adverse events as soon as possible, but no later than 24 hours after becoming aware of the event;
- Adhere to the publication policy, as stated in the Clinical Study Agreement, for data collected during this study; and
- Ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

I will ensure that the Institutional Review Board (IRB) / Ethics Committee (EC) review complies with governmental requirements and will be responsible for the initial and continuing review and approval of the clinical investigation. I also agree to promptly report to the IRB/EC all changes in the research activity and all unanticipated problems involving risks to human subjects or others. Additionally, I will not make any changes in the research without sponsor and IRB/EC approval of an amended protocol, except where necessary to eliminate apparent immediate hazards to human subjects.

I agree to comply with all other requirements regarding the obligation of clinical investigators and all other pertinent requirements of the sponsor and government agencies.

| Investigator Signature | Date |
|------------------------------|----------|
| | <u>-</u> |
| Printed Name of Investigator | |



# **SYNOPSIS**

| Regulatory<br>Classification: | Class II Staple Implantable; Stapler, Surgical 21CFR 878.4750. Cleared 11/24/2014, 510(k) # K141952 |
|---|---|
| | CE Mark granted 02/27/2015, Certificate, G7 15 02 57666 049 |
| Indication: | The ECHELON FLEX <sup>™</sup> Powered Vascular Stapler (PVS) with Advanced Placement Tip and its reloads are intended for transection and resection of tissue and vasculature. The instruments have application in multiple open or minimally invasive general, gynecologic, urologic, thoracic, and pediatric surgical procedures. The device will be utilized as described in the instruction for use (IFU). |



# Objective/Primary Endpoints:

The primary objective of the trial is to demonstrate that the frequency of hemostatic interventions/procedures required intra-operatively or post-operatively related to the transection of the renal artery (RA) and renal vein (RV) during laparoscopic nephrectomies and nephroureterectomies with powered vascular stapler (PVS) is not increased when compared to standard of care (SOC).

The primary performance endpoint will be:

Incidence of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the RA and RV during laparoscopic nephrectomies and nephroureterectomies with the use of standard of care stapler (SOC) or powered vascular stapler (PVS) defined as:

 Hemostasis intervention: bleeding detected and controlled intra-operatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intraoperatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).

No hemostasis intervention is defined as no bleeding at the staple line or bleeding that stops after initial blotting of staple line.

The primary safety endpoint will be:

Incidence of hemostatic interventions /procedures completed for post-operative bleeding related to the transection of the RA and RV during during laparoscopic nephrectomies and nephroureterectomies with the use of SOC or PVS:

 Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to RA and RV transection).

No hemostasis intervention is defined as no interventions needed for post-operative bleeding (related to RA and RV transection).



| Study Design: | This prospective, randomized, controlled, multi-center study will collect and compare data from the surgeon's current SOC stapler (for RA/RV transection) and powered vascular stapler. |
|---|---|
| Number of<br>Subjects<br>(Planned): | Approximately 250 subjects will be randomized |
| Diagnosis/Criteria for Inclusion: | Subjects satisfying the following criteria will be eligible for participation in this study: |
| | <ol> <li>Scheduled for a simple or radical laparoscopic nephrectomy or a laparoscopic nephroureterectomy in accordance with the institution's standard of care (SOC);</li> <li>Performance status 0-1 (Eastern Cooperative Oncology Group classification), if applicable;</li> <li>ASA score ≤ 3;</li> <li>No prior history of partial or wedge nephrectomy (on the kidney in which the procedure will be performed);</li> <li>Willing to give consent and comply with study-related evaluation and treatment schedule; and</li> <li>At least 18 years of age.</li> </ol> |
| Diagnosis/Criteria for Exclusion: | Subjects will be excluded from the study for any of the following: 1. Prior chemotherapy or radiation (within 30 days prior to the procedure or the duration of the subject's enrollment); |
| | <ol> <li>Pregnancy;</li> <li>Physical or psychological condition which would impair study participation; or</li> <li>The subject is judged unsuitable for study participation by the Investigator for any other reason.</li> </ol> |
| Finished Product: | ECHELON FLEX <sup>™</sup> Powered Vascular Stapler with Advanced Placement Tip |



# Statistical Methods:

Summary statistics and 95% confidence intervals will be provided for the number and frequency of interventions for the set of SOC and PVS subjects separately. This will be performed based on the total number of firings. An intervention is defined as any firing which is classified as hemostasis intervention. Given that it is expected to have at least 300 firings in each group, the sample size of approximately 250 subjects is considered adequate for descriptive summarization of the number and frequency of surgical interventions. Assuming an approximate background intervention rate of 6%, the given sample size will provide reasonable precision in the estimation of the intervention rate to an expected margin of error for a 95% confidence interval of at most 2.9% for each group. To establish that the intervention rate is not increased compared to SOC, a 95% confidence interval for the difference in proportion of firings requiring interventions for PVS minus SOC will be calculated and powered vascular stapler will be considered to have acceptable performance if the upper bound of the 95% confidence interval does not exceed 3%.

The number and percentage of subjects requiring hemostasis interventions post-operatively that are classified as related to SOC or PVS for RA/RV transection (e.g. need for blood product transfusion or additional surgical procedure) will be summarized for each group as a primary safety endpoint.

Additional endpoints will be summarized with descriptive statistics and 95% confidence intervals as appropriate for continuous or categorical measurements

Safety will be assessed through the incidence of AEs and serious adverse events (SAEs), which will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).



# **SCHEDULE OF EVENTS**

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| Study Activity | Screening | Procedure | Post-Op<br>through<br>Discharge | 4 week<br>followup <sup>d</sup><br>(post<br>procedure) |
| Informed consent | X | | | |
| Demographic information | X | | | |
| Relevant medical/surgical history | X | X | | |
| Inclusion/Exclusion Criteria | X | X | | |
| ASA score | | X | | |
| Randomization (SOC or PVS) | | Х | | |
| Collection of procedure data <sup>a</sup> | | Х | | |
| Intra-operative interventions on RA/RV | | Х | | |
| Post-operative interventionson on RA/RV | | | Х | Х |
| Procedure duration | | Х | | |
| Device usage data | | X | | |
| Daily volume and characteristics of drainage (drains) | | | Х | X |
| Concomitant Procedures/interventions, if applicable | | | Х | Х |
| Surgeon questionnaires <sup>b</sup> | | Х | | |
| Date of hospital admission | | X | | |
| Overall Operating Room (OR) time | | Х | | |
| Adverse Events | | Х | Х | Х |
| Anticoagulants <sup>c</sup> | X | | | |
| Concomitant medications associated with adverse events | | X | Х | X |
| Date of drain removal, if applicable | | | Х | Χ |
| Discharge date | | | Х | |
| Subject exited from study | | | | X |

a. See section 4.7.3.2 for specific details
 b. Surgeon Device Questionnaire (*PVS procedures only*). Surgeon Satisfaction and SURG-TLX (*SOC and PVS procedures*)
 c. Anticoagulants taken preoperatively (up to 30 days prior to Visit 2), including the stop date
 d. Phone call or office visit



# **TABLE OF CONTENTS**

| | Page |
|----------------------------------------------------------------|-----------|
| INVESTIGATOR SIGNATURE | 3 |
| SYNOPSIS | |
| SCHEDULE OF EVENTS | 8 |
| ETHICS | |
| ADMINISTRATIVE REQUIREMENTS | 12 |
| 1.0 INTRODUCTION AND BACKGROUND | |
| 2.0 STUDY OBJECTIVES | |
| 2.1 PRIMARY OBJECTIVE | 14 |
| 3.0 INVESTIGATIONAL PLAN | |
| 3.1 GENERAL DESIGN | |
| 3.2 PRIMARY ENDPOINTS | 14 |
| 3.3 ADDITIONAL MEASUREMENTS / DATA COLLECTED | 15 |
| 4.0 INVESTIGATIONAL PLAN | 15 |
| 4.1 OVERALL STUDY DESIGN | 15 |
| 4.2 RANDOMIZATION | 16 |
| 4.2.1 INCLUSION CRITERIA | |
| 4.2.2 EXCLUSION CRITERIA | 16 |
| 4.3 PRIOR AND CONCOMITANT THERAPY | |
| 4.3.1 CONCOMITANT MEDICATIONS | |
| 4.4 REMOVAL OF SUBJECTS FROM STUDY | |
| 4.5 IDENTITY OF STUDY PRODUCT(S) | 18 |
| 4.6 PRODUCT ACCOUNTABILITY | |
| 4.7 STUDY PROCEDURES | |
| 4.7.1 PROCEDURE DESCRIPTION | 19 |
| 4.7.2 VISIT 1 – SCREENING (CAN OCCUR OVER SEVERAL DATES WITHIN | 1-2 WEEKS |
| OF VISIT 2- PROCEDURE) | |
| 4.7.3 VISIT 2 –PROCEDURE | |
| 4.7.3.1 PRE-PROCEDURE | |
| 4.7.3.2 INTRAOPERATIVE | |
| 4.7.4 VISIT 3 – POSTOPERATIVE THROUGH DISCHARGE | |
| 4.7.5 VISIT 4-FINAL VISIT (4 WEEK FOLLOW UP, POST PROCEDURE) | |
| 5.0 DATA MANAGEMENT AND INTEGRITY | |
| 5.1 DATA COMPLETION AND RECORD KEEPING | |
| 5.1.1 Source Documents | |
| 5.1.2 Electronic Data Capture | |
| 5.1.3 Data Collection | |
| 5.1.4 Data Correction | |
| 5.1.5 Data Privacy | |
| 5.1.6 Record Retention, Inspection, and Custody | ∠3 |



| 5.2 | MEDICAL DICTIONARY CODING | 23 |
|---|---|---|
| 6.0 | DATA QUALITY ASSURANCE | 23 |
| 6.1 | INVESTIGATOR TRAINING | 23 |
| 6.2 | MONITORING | |
| 6.3 | PROTOCOL DEVIATIONS | 24 |
| 7.0 | STATISTICAL METHODS PLANNED IN THE PROTOCOL AND DETERMINATION | OF |
| SAMF | PLE SIZE | |
| 7.1 | STATISTICAL AND ANALYTICAL PLANS | 24 |
| 7.2 | DETERMINATION OF SAMPLE SIZE | 24 |
| 7.3 | ANALYSIS SETS | 24 |
| 7.4 | ANALYSIS OF EFFECTIVENESS | |
| 7.5 | STATISTICAL/ANALYTICAL ISSUES | |
| 7.5.1 | HANDLING OF DROPOUTS OR MISSING DATA | |
| 7.5.2 | INTERIM ANALYSES AND DATA MONITORING | |
| 7.5.3 | MULTICENTER STUDIES | |
| 7.5.4 | MULTIPLE COMPARISONS/MULTIPLICITY | |
| 7.6 | ANALYSIS OF SAFETY | 25 |
| 8.0 | RISKS AND BENEFITS OF THE STUDY DEVICE AND CLINICAL INVESTIGATION | |
| 9.0 | ADVERSE EVENTS AND PRODUCT COMPLAINTS | |
| 9.1 | DEFINITIONS | |
| 9.1.1 | ADVERSE EVENT | |
| 9.1.2 | ANTICIPATED ADVERSE EVENTS | |
| 9.1.3 | SERIOUS ADVERSE EVENT | |
| 9.1.4 | SEVERITY OF ADVERSE EVENTS | |
| 9.1.5 | RELATIONSHIP OF ADVERSE EVENTS | |
| 9.1.6 | PRODUCT COMPLAINTS | |
| 9.2 | REPORTING PROCEDURES FOR ADVERSE EVENTS/PRODUCT COMPLAINTS | 28 |
| | 28 | |
| 9.2.1 | REPORTING ADVERSE EVENTS | |
| 9.2.2 | REPORTING SERIOUS ADVERSE EVENTS | |
| 9.2.3 | REPORTING PRODUCT COMPLAINTS | _ |
| 10.0 | REFERENCE LIST | 29 |
| APPE | ENDIX I: ANTICIPATED ADVERSE EVENTS | 30 |



## **ETHICS**

#### **Institutional Review Board/Ethics Committee**

Participating investigators will ensure that this protocol, Informed Consent Document (ICD), ICD or protocol amendments, and if applicable, any other written information provided to the subjects that assist in the decision to participate are reviewed by an Institutional Review Board (IRB) or Ethics Committee (EC) that complies with governmental requirements. The approving IRB/EC will be responsible for the initial and continuing review and approval of this clinical investigation. Participating investigators will be required to promptly report to the IRB/EC as required by the IRB/EC's policies. Additionally, investigators will be required to refrain from making any changes in the clinical investigation plan without Sponsor and IRB/EC approval of an amended protocol, except where necessary to eliminate apparent immediate hazards to study subjects or others.

# Applicable Regulations

This study will be conducted in compliance with Good Clinical Practice and in accordance with the Declaration of Helsinki, ISO 14155:2011, as well as any other applicable local and country regulatory requirements.

## **Subject Information and Consent**

Regulations concerning the protection of subjects require that informed consent be obtained before a subject may participate in any clinical investigation.

An IRB/EC approved informed consent must be sought from each subject and must be appropriately documented in the subject's medical record prior to initiating the study. It is the Investigator's responsibility to obtain written informed consent from the subject. The Investigator may delegate this responsibility if appropriately documented.

The informed consent process involves the following: giving a subject adequate information concerning the study, providing adequate time for the subject to consider all available options. responding to the subject's questions, ensuring that the subject has comprehended this information and finally, obtaining the subject's written consent to participate in this study. All subjects in this study should be completely informed about the purpose, risks, benefits, and other pertinent details of this study. The informed consent process is careful to avoid the perception of any coercion or undue influence on, or inducement of, the subject to participate, and does not waive or appear to waive the subject's legal rights. The ICD is presented in native, non-technical language that is understandable to the subject.

Prior to a subject's participation in this study, an ICD will be signed and dated by the subject and person who conducted the consent discussion. The subject will be provided a copy of the signed ICD. The ICD and any other written materials provided to the subject to assist in the decision to participate must be revised whenever new information becomes available that may be relevant to their willingness to participate or continue participation in this study. Revision to the ICD and other written materials will receive IRB/EC approval before implementation. Each subject will be required to sign any amended ICD (as required by the IRB/EC) and will receive a copy of the signed ICD.

CONFIDENTIAL Protocol ESC-15-002 



## ADMINISTRATIVE REQUIREMENTS

This study is sponsored by Ethicon Endo-Surgery, Inc. (EES, Cincinnati, OH, USA) and will be conducted in approximately eight surgery centers in the United States and/or European Union under a single protocol approved by each participating site's IRB/EC prior to implementation. The principal investigator at each study site is a surgeon qualified by education, experience, and training to perform the study procedure and to assume responsibility for the conduct of this study.

The Data Management and Biostatistics groups of Ethicon Endo-Surgery, Inc.'s Global Surgery Clinical Development will be responsible for the analysis of data from this protocol. An Electronic Data Capture (EDC) system will be utilized by study site personnel to transfer study data from source records (the first point of clinical data capture) onto common electronic case report forms (eCRFs). This system is a web-based, secure electronic software application (Medidata® Rave, 350 Hudson Street, 9th Floor, New York, New York, 10014). This system was designed and is developed and maintained by Medidata in a manner that is compliant with national and international Good Clinical Practice (GCP) data protection/data privacy and electronic record/electronic signature (e.g. 21 CFR Part 11) regulatory requirements.

#### **Protocol Modifications**

All protocol amendments must be issued by the Sponsor, signed and dated by the Investigator, and should not be implemented without prior IRB/EC only logistical or administrative aspects of the study (e.g., change in Sponsor personnel, change of telephone number(s)). The Investigator will submit the protocol amendments to the IRB approval, except where necessary to eliminate immediate hazards to the subjects or when the change(s) involves /EC as per their local requirements.



## 1.0 INTRODUCTION AND BACKGROUND

Nephrectomy has many indications, for both simple and radical approaches. A simple nephrectomy is indicated in patients with irreversible kidney damage due to symptomatic chronic infection, obstruction, calculus disease, or severe traumatic injury. Simple nephrectomy is also indicated to treat renovascular hypertension due to noncorrectable renal artery disease or severe unilateral parenchymal damage caused by nephrosclerosis, pyelonephritis, reflux dysplasia, or congenital dysplasia of the kidney. <sup>1</sup>

Surgery (traditional or laparoscopic) is the primary treatment for most renal cancers<sup>2</sup> while laparoscopic donor nephrectomy has remained a safe, less invasive, and effective technique for renal allograft procurement.<sup>3</sup>

The most common reason for a nephroureterectomy (removal of the kidney and ureter) is transitional cell carcinoma. Transitional cell carcinoma is a cancer that occurs within the transitional epithelium of the kidney, ureter, and/or bladder.

The surgical procedures performed under this protocol are simple or radical laparoscopic nephrectomies or nephroureterectomies. The laparoscopic approach typically utilizes several small incisions in the abdominal and/or flank area. Through these incisions, a surgeon uses a camera and specialized surgical instruments to conduct the operation and remove the entire affected kidney (and some of the surrounding tissues if indicated). Laparoscopic nephrectomy is associated with less postoperative pain and a faster return to normal activities than open nephrectomy.<sup>4</sup>

The ECHELON FLEX<sup>™</sup> Powered Vascular Stapler with Advanced Placement Tip can transect vessels in restricted narrow spaces near delicate vascular anatomy. With its narrow anvil and curved dissection tip, this stapler enhances visibility and provides precise placement.

Protocol ESC-15-002  Version/Date: Original/17 NOV2015 FINAL



#### 2.0 STUDY OBJECTIVES

#### 2.1 PRIMARY OBJECTIVE

The primary objective of the study is to demonstrate that the frequency of hemostatic interventions/procedures required intra-operatively or post-operatively related to the transection of the renal artery (RA) and renal vein (RV) during simple, radical laparoscopic nephrectomies or laparoscopic nephroureterectomies with PVS is not increased when compared to standard of care (SOC).

#### 3.0 INVESTIGATIONAL PLAN

#### 3.1 GENERAL DESIGN

This prospective, randomized, controlled, multi-center study will collect and compare data from the surgeon's current SOC stapler (for RA/RV transection) and PVS. Approximately 250 individuals undergoing simple or radical laparoscopic nephrectomies or laparoscopic nephroureterectomies, and who meet study entry criteria, will be randomized in a 1:1 ratio to either the surgeon's current SOC stapler or PVS. Prospective subjects will be informed about the nature of the research, given the ICD to read, and if the subject understands the consent, will be asked to provide written consent (the ICD).

#### 3.2 PRIMARY ENDPOINTS

The primary performance endpoint will be:

Incidence of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the RA and RV during laparoscopic nephrectomies and nephroureterectomies with the use of standard of care stapler (SOC) or powered vascular stapler (PVS) defined as:

 Hemostasis intervention: bleeding detected and controlled intra-operatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).

No hemostasis intervention is defined as no bleeding at the staple line or bleeding that stops after initial blotting of staple line.

The primary safety endpoint will be:

Incidence of hemostatic interventions /procedures completed for post-operative bleeding related to the transection of the RA and RV during laparoscopic nephrectomies and nephroureterectomies with the use of SOC or PVS:

 Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to RA and RV transection).

Protocol ESC-15-002 Version/Date: Original/17 NOV2015 FINAL



No hemostasis intervention is defined as no interventions needed for post-operative bleeding (related to RA and RV transection).

#### 3.3 ADDITIONAL MEASUREMENTS / DATA COLLECTED

- a. Subject demographics;
- b. All adverse events:
- c. Anticoagulants taken preoperatively (up to 30 days prior to Visit 2) and concomitant medications associated with AEs;
- d. Relevant medical/surgical history (including hypertension, if applicable);
- e. Procedure details:
- f. Number of ports;
- g. Overall operating room and procedure duration;
- h. Intraoperative and postoperative surgical interventions (not associated with transection of the RA/RV), if applicable;
- i. Volume of estimated intra-operative blood loss;
- j. Date(s) of drain removal;
- k. Daily volume and characteristics of drainage;
- Transfusion of blood or blood products;
- m. Device usability /articulation questions;
- n. Surgeon assessment of visualization;
- o. Surgeon Questionnaires;
- p. Concomitant procedures/interventions, if applicable; and
- q. Length of stay (LOS) from admission through discharge.

The data collected for this study may be used for future research or enhancement of similar surgical tools.

#### 4.0 INVESTIGATIONAL PLAN

## 4.1 OVERALL STUDY DESIGN

This is a prospective, randomized, controlled, multi-center study that is intended to demonstrate that the frequency of hemostatic interventions/procedures required intra-operatively or post-operatively related to the transection of the renal artery (RA) and renal vein (RV) during simple, radical laparoscopic nephrectomies or laparoscopic nephroureterectomies with PVS is not increased when compared to standard of care (SOC).

Eligible subjects will be randomized pre procedure in a 1:1 ratio to either the surgeon's current SOC stapler or PVS. Subjects will be followed post-operatively through discharge and at 4 weeks post surgery (final visit can be conducted either by phone or office visit).

If the study surgeons have not completed previous ECHELON FLEX<sup>TM</sup> Powered Vascular Stapler with Advanced Placement Tip training, each surgeon must complete two procedures with ECHELON FLEX<sup>TM</sup> Powered Vascular Stapler with Advanced Placement Tip prior to their first randomized subject. These subjects will be considered part of a learning curve and will be analyzed separately from the randomized subjects.

Protocol ESC-15-002 

Version/Date: Original/17 NOV2015 FINAL



#### 4.2 RANDOMIZATION

In this non blinded study, randomization will be used to avoid bias in the assignment of the stapling device to be utilized for RA/RV transection for each subject, to increase the likelihood that attributes of the subject are evenly balanced between groups, and to enhance the validity of statistical comparisons between groups.

The Sponsor will assign the stapling device randomly to each subject on a 1:1 basis to either the surgeon's current SOC or PVS.

In the event that a potential subject fails inclusion/exclusion criteria prior to randomization, this subject will be considered a screen failure.

#### 4.2.1 Inclusion Criteria

Subjects satisfying the following criteria will be eligible for participation in this study:

- 1. Scheduled for a simple or radical laparoscopic nephrectomy or a laparoscopic nephroureterectomy in accordance with the institution's standard of care (SOC);
- 2. Performance status 0-1 (Eastern Cooperative Oncology Group classification), if applicable;
- 3. ASA score  $\leq$  3;
- 4. No prior history of partial or wedge nephrectomy (on the kidney in which the procedure will be performed);
- 5. Willing to give consent and comply with study-related evaluation and treatment schedule; and
- 6. At least 18 years of age.

#### 4.2.2 Exclusion Criteria

Subjects will be excluded from the study for any of the following:

- 1. Prior chemotherapy or radiation (within 30 days prior to the procedure or the duration of the subject's enrollment);
- 2. Pregnancy;
- 3. Physical or psychological condition which would impair study participation; or
- 4. The subject is judged unsuitable for study participation by the Investigator for any other reason

All subjects signing consent who do not meet the inclusion/exclusion criteria and therefore do not proceed to Visit 2/Procedure, and are not randomized, will be recorded as screen failures. The relevant electronic Case Report Form (eCRF) pages will be completed for all screen failure subjects and the data will therefore be included in the study database.

#### 4.3 PRIOR AND CONCOMITANT THERAPY

Study subjects may continue with their current medical care while in the study, including medications.

Protocol ESC-15-002 



#### 4.3.1 Concomitant Medications

Anticoagulants taken preoperatively (up to 30 days prior to Visit 2) and medications prescribed due to an adverse event will be collected for this study. No other concomitant medications will be collected.

### 4.4 REMOVAL OF SUBJECTS FROM STUDY

A subject has the right to withdraw from the study at any time for any reason without prejudice to his/her future medical care by the physician or the institution. Should a subject (or subject's legally authorized guardian/representative) decide to withdraw; all efforts will be made to collect and report the final visit observations as thoroughly and timely as possible.

Subjects who withdraw from the study prior to randomization will be considered screen failures and will be replaced. Subjects who withdraw from the study post-randomization, will not be replaced. Subject participation may be terminated prior to completing the study for any of the reasons listed below. When a subject's participation is terminated prior to completing the study, the reason for withdrawal is to be documented on the Study Completion eCRF as well as in the source documentation:

#### Withdrawal of Consent:

The subject withdraws consent for participation in the study. Any method of contact with the subject in which they state they no longer want to participate in the study specific activities constitutes withdrawal of consent. When possible the reason for withdrawal of consent will be documented.

#### Surgical:

The Investigator must withdraw a subject intraoperative for the following reasons:

- A simple or radical laparoscopic nephrectomy or laparoscopic nephroureterectomy not completed;
- Conversion to an open procedure, unless directly related to transection of the RA/RV (subject will be followed for safety up to 30 days postop); or
- Use of robotic assistance during surgery.

#### Adverse Event:

 When the subject experiences an adverse event and the Principal Investigator or Medical Director believes it is in their best interest to discontinue participation in the study, they will be withdrawn.

## Death:

When possible, the cause of death will be documented.

# Lost to follow-up:

When contact with the subject has been lost without completing a final visit assessment, and every attempt to contact has failed, the subject will be considered lost to follow-up. Final

Protocol ESC-15-002 

Version/Date: Original/17 NOV2015 FINAL



documentation regarding all attempts to contact the subject requesting their return for the final visit should be documented.

#### Site Termination or Study Termination:

A site or study may be terminated. When this occurs all subjects at the site will be withdrawn and documented as early termination. Reasons for site or study termination may include, but are not limited to the following:

- Administrative Concerns (e.g., inadequate subject enrollment, investigator/institution non-compliance, change of business strategy, etc.);
- Safety Issues, including those due to non-compliance, which substantially affect the risk to benefit ratio of the study subjects at a site or for the study as a whole; and
- Regulatory Body Mandate(s).

The Investigator has the right to terminate their participation at any time. Should this be necessary, procedures for termination will be provided by the Sponsor.

# 4.5 IDENTITY OF STUDY PRODUCT(S)

| Product<br>Code | Product Name | Manufacturer |
|---|---|---|
| PVE35A | ECHELON FLEX™ Powered Vascular Stapler with Advanced Placement Tip | Ethicon Endo-Surgery,<br>LLC (Guaynabo, Puerto<br>Rico, USA) |
| VASECR35 | ENDOPATH ECHELON Vascular White Reload for Advanced Placement Tip | Ethicon Endo-Surgery,<br>LLC (Guaynabo, Puerto<br>Rico, USA) |

The ECHELON FLEX™ Powered Vascular Stapler with Advanced Placement Tip is a sterile, single use instrument that simultaneously cuts and staples tissue. There are four staggered rows of staples, two on either side of the cut line. The ECHELON FLEX™ Powered Vascular Stapler with Advanced Placement Tip and reloads have a staple line that is approximately 35mm long and a cut line that is approximately 30 mm long. The shaft can rotate freely in both directions and an articulation mechanism enables the distal portion of the shaft to pivot to facilitate lateral access to the operative site.

Powered vascular stapler has been cleared for marketing by the FDA and is CE marked which allows for commercial distribution in the EU. The device will be used in accordance with product labeling and Instructions for Use (IFU).

# 4.6 PRODUCT ACCOUNTABILITY

The ECHELON FLEX™ Powered Vascular Stapler with Advanced Placement Tip and cartridges will be provided by the Sponsor and will be tracked using shipping invoices and device accountability logs. All product returns will be managed by contacting the Sponsor.

Protocol ESC-15-002 



The powered vascular staplers must be kept in a secure area. Devices will only be used for treating subjects participating in the study, in accordance with the protocol. The study device inventory must be available for periodic inspection/verification.

#### 4.7 STUDY PROCEDURES

# 4.7.1 Procedure Description

A simple or radical laparoscopic nephrectomy or a laparoscopic nephroureterectomy will be performed according to the institution's SOC.

# 4.7.2 Visit 1 – Screening (can occur over several dates within 1-2 weeks of Visit 2- Procedure)

Subjects will be evaluated according to the local investigator's preferred practice. Subjects will be selected for a surgical procedure based on the preoperative investigations and the local investigator's interpretation of the clinical picture.

Eligible subjects will be provided with the study information including the ICD.

The following screening activities will occur prior to the study procedure:

- The subject must be given ample time to review and sign the ICD;
- Collection of demographic information (year of birth, gender, ethnicity);
- Review and collection of relevant medical/surgical history, history of hypertension if applicable;
- Review/collection of inclusion/exclusion criteria and determination as to whether
  the subject is eligible for participation (retrospective data, per site SOC, is
  permitted to determine eligibility); and
- Anticoagulants taken preoperatively (up to 30 days prior to Visit 2), including stop date

#### 4.7.3 Visit 2 - Procedure

#### 4.7.3.1 Pre-procedure

The following must be obtained prior to the surgical procedure:

- Date of hospital admission;
- Update to medical / surgical history, if applicable;
- Confirm inclusion and exclusion criteria;
- ASA score; and
- Randomization

# 4.7.3.2 Intraoperative

Data collected during procedure:

• Overall Operating Room (OR) time;

Protocol ESC-15-002  Version/Date: Original/17 NOV2015 FINAL



- Duration of procedure (first incision to skin closure);
  - Includes time to completion of resection (capturing the time laparoscopic camera is inserted until the specimen is received)
- Procedure data:
  - Type of surgery;
  - Number of renal arteries (1, 2, or 3+);
  - Location of affected kidney;
  - Confirm visualization of the cut line indicator field prior to transection;
  - Number of ports;
  - Intraoperative surgical interventions (not associated with transection of the RA/RV), if applicable;
  - Number and type of drain tubes placed, if applicable;
  - Reason for conversion to open surgery, if applicable;
  - Volume of estimated intra-operative blood loss;
  - Transfusion products (and rationale for use), if applicable;
  - Concomitant procedures/interventions performed, if applicable;
  - Tumor size and TNM staging, if available or applicable
- Intra-operative interventions/procedures on RA/RV to stop bleeding, if applicable;
  - Hemostasis intervention: bleeding detected and controlled intraoperatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).
- Device usage data:
  - Usability and articulation questions;
- Surgeon Device Questionnaire (PVS procedures only);
- Surgeon Satisfaction Questionnaire (SOC and PVS procedures);
- SURG-TLX (SOC and PVS procedures);
- Adverse Events; and
- Concomitant medication (associated with AEs)

# 4.7.4 Visit 3 – Postoperative through Discharge

Post procedure assessments will be completed from OR discharge until hospital discharge. Data to be collected includes:

 Post-operative interventions/procedures related to RA/RV bleeding, if applicable:

Protocol ESC-15-002 



- Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (and the relationship to SOC/PVS for RA/RV transection);
- Date of drain removal, if applicable
- Daily volume and characteristics of drainage (drain);
- Concomitant procedures/ interventions performed, if applicable;
- Adverse Events;
- Concomitant medication (associated with AEs); and
- Discharge date

# 4.7.5 Visit 4-Final Visit (4 week follow up, post procedure)

This visit can be either an office visit or a telephone followup visit. Data to be collected includes:

- Post-operative interventions/procedures related to RA/RV bleeding, if applicable:
  - Hemostasis intervention: Bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (and the relationship to SOC/PVS for RA/RV transection);
  - Concomitant procedures/interventions performed, if applicable;
  - Date of drain removal, if applicable
  - Daily volume and characteristics of drainage (drain), if applicable;
  - Adverse Events;
  - Concomitant medication (associated with AEs); and
  - Subject exited from the study

#### 5.0 DATA MANAGEMENT AND INTEGRITY

#### 5.1 DATA COMPLETION AND RECORD KEEPING

#### 5.1.1 Source Documents

Source documents are documents on which information regarding subjects is first recorded, including printed, hand written, or electronic documents. Investigator subject files or hospital records generally are the basis of source document information. This includes but is not limited to, original subject files; hospital/clinic records; original recordings /tracing; digital images from automated instruments (e.g., cameras); radiographs; device accountability records; photographic negatives; and records kept at the investigation site, at the laboratories and at other departments involved in the clinical investigation.

Source documents must be retained by the Investigator as part of the subject's permanent medical record. The information in the source documents is used to complete the eCRFs. All information captured on the eCRFs should be completely and accurately supported in source documentation. Any additional

Protocol ESC-15-002 Version/Date: Original/17 NOV2015 FINAL



information relevant to the study should be included in the source documents. The Investigator will retain originals of all source documents, subject consent forms, and study data.

# **5.1.2** Electronic Data Capture

An electronic data capture (EDC) system will be utilized by study site personnel to transfer study data from source records (medical records and/or source document worksheets) onto common eCRFs. This system is a web-based, secure electronic software application (Medidata® Rave, Medidata® Rave, 350 Hudson Street, 9th Floor, New York, New York, 10014). This system was designed and is developed and maintained by Medidata in a manner that is compliant with national and international GCP data protection/data privacy and electronic record/electronic signature (e.g., 21 CFR Part 11) regulatory requirements. The EDC system will be used to facilitate the collection of all study data at the site. Designated site personnel will be responsible for entering subject data into the EDC system. All external and Sponsor internal users will be trained on the EDC application at a level dependent on their planned function. An EDC digital User Manual will be available under the help menu within the Medidata® Rave website to assist in the collection and entry of source data into the electronic casebook.

There is a 24/7/365 Help Desk Support line staffed by the outsourced vendor that will be available to respond to questions.

#### 5.1.3 Data Collection

Each EDC eCRF will be completed by the PI or PI's designee. Every effort should be made to respond to all monitoring and/or data management questions on each eCRF as completion of the data is required by the protocol. A unique ID number will identify each subject. The subject's unique ID number will be visible on each eCRF. At no time should the subject name appear on the eCRFs.

All data should be recorded accurately and completely. The Investigator is responsible for reviewing and approving each completed eCRF. Assurance of overall review and approval will be documented by the Investigator electronically signing each subject's electronic casebook.

#### 5.1.4 Data Correction

Required data corrections to eCRFs will be prompted via automated electronic edit checks and/or queries manually created by Sponsor reviewers. The change(s), individual making the change(s), and time the change(s) were made to the eCRFs will be automatically captured in the audit trail within Medidata<sup>®</sup> Rave.

# 5.1.5 Data Privacy

The collection, use, and disclosure of all personal data, including subject health and medical information, are to be maintained in compliance with applicable personal data protection and security laws and regulations that govern protected health information and the informed consent given by each study subject. When collecting and processing such personal data, appropriate measures are to be taken to maintain the confidentiality of subject health and medical information and



to prevent access by unauthorized persons.

# 5.1.6 Record Retention, Inspection, and Custody

The PI must maintain all documentation related to the study until they receive Sponsor notification. The PI will allow representatives of the Sponsor, the FDA, or other applicable government regulatory agencies to inspect all study records, eCRFs, and corresponding portions of the subject's office and/or hospital medical records at regular intervals during the study. These inspections are to verify adherence to the protocol, integrity of the data being captured on the eCRFs, and compliance with applicable regulations.

Subject medical records will be maintained in a confidential manner. Study reports will not identify subjects by name. These reports may be submitted to the FDA and/or applicable regulatory authorities.

If custody of the records is transferred, notice of such a transfer should be given to the Sponsor no later than 10 working days after the transfer occurs.

#### 5.2 MEDICAL DICTIONARY CODING

Medical dictionary coding of verbatim AE, and SAE captured on eCRFs will be performed using a coding thesaurus algorithm. The Medical Dictionary for Regulatory Activities and World Health Organization Drug Dictionary will be used after data entry and query resolution, via auto-encoding and interactive coding processes.

#### 6.0 DATA QUALITY ASSURANCE

Steps to be taken to assure the accuracy and reliability of data include the selection of qualified investigators and appropriate study centers, review of protocol procedures with the Investigator and associated personnel prior to the study, and periodic monitoring visits by the Sponsor. The Sponsor will review eCRFs for accuracy and completeness during on-site monitoring visits or periodic reviews of the EDC system; any discrepancies will be resolved with the Investigator or designees, as appropriate. The data entered into the clinical study database will be verified for accuracy.

## **6.1 INVESTIGATOR TRAINING**

Prior to screening subjects for this study, the PI, sub-investigators, study coordinators, and other designated staff (as applicable) will be provided information on study execution, data collection, and procedures specific to this clinical protocol.

#### 6.2 MONITORING

This study will be monitored by the Sponsor to ensure:

- The rights and well-being of the subjects are protected;
- Reported study data is accurate, complete, and verifiable from source documents; and
- The conduct of the study is in compliance with the currently approved protocol/amendment(s), applicable GCPs, and with applicable local/regional regulatory requirements.

The extent and nature of monitoring will be predetermined and based on considerations

Protocol ESC-15-002 CONFIDENTIAL
Version/Date: Original/17 NOV2015 FINAL



such as the objective, design, complexity, and endpoints of the study and mutually agreed to by the Sponsor and investigators. Monitors will comply with established written standard operating procedures as well as procedures (i.e., monitoring plan) specified by the Sponsor for monitoring this study. These monitoring procedures are characterized in the monitoring plan for this study.

#### 6.3 PROTOCOL DEVIATIONS

A deviation (any activity conducted outside the parameters established by the study protocol) can be identified from a number of sources. Potential sources include, but are not limited to: a member of the Investigator's staff, a Sponsor representative during monitoring visits, or a member of the data management or statistical groups when entering or analyzing data. Regardless of the source, it is crucial to document the deviation. The PI will report protocol deviations to the IRB/EC as required by the IRB/EC procedures. All deviations will be captured in the source as well as the eCRF.

# 7.0 STATISTICAL METHODS PLANNED IN THE PROTOCOL AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL AND ANALYTICAL PLANS

The Sponsor's Data Management and Biostatistics groups will be responsible for the analysis of data from this protocol. A comprehensive and detailed Statistical Analysis Plan (SAP) will be finalized prior to database lock and will supplement the statistical design and analysis described in this section.

Categorical variables will be summarized descriptively by frequencies and associated percentages. Continuous variables will be summarized descriptively by number of subjects, mean, standard deviation, median, minimum, and maximum.

# 7.2 DETERMINATION OF SAMPLE SIZE

Approximately 250 subjects will be randomized in the study in a 1:1 ratio to standard of care or powered vascular stapler. Historical clinical study data on a similar powered surgical stapler demonstrated a need for staple line interventions in approximately 6% of firings on the pulmonary artery or pulmonary vein. This data also showed an average of 2.6 to 2.9 firings per subject, and it is expected, given differences in device design and procedure, that each subject will require 2 to 3 firings on the renal vein or renal artery in the current study with powered vascular stapler.

Given that it is expected to have a minimum of 300 firings in each group, the sample size of approximately 250 subjects is considered adequate for descriptive summarization of the primary performance endpoint, i.e. number and frequency of intra-operative surgical interventions. Assuming an approximate background intervention rate of 6%, the given sample size will provide reasonable precision in the estimation of the intervention rate to an expected margin of error for a 95% confidence interval of at most 2.9% for each group.

#### 7.3 ANALYSIS SETS

There will be three analysis sets defined:

• The Full Analysis Set (FAS) will consist of all randomized subjects who had the

Protocol ESC-15-002 Version/Date: Original/17 NOV2015 FINAL



procedure performed and provide data on number of surgical interventions;

- The Per Protocol (PP) Analysis Set will consist of all subjects in the FAS who had no major protocol violations;
- The Safety Set consists of all randomized subjects on whom the procedure is started.

The primary performance endpoint analysis will be performed on the Full Analysis Set and subjects will be classified according to their randomized treatment group. The primary endpoint analysis will also be performed on the PP set as a sensitivity analysis to the results on the FAS. The summary of additional endpoints will also be performed on the Full Analysis Set. Analysis of the primary safety endpoint and adverse event summaries will be performed on the Safety Set.

## 7.4 ANALYSIS OF EFFECTIVENESS

Summary statistics and 95% confidence intervals will be provided for the number and frequency of interventions for the set of SOC subjects and PVS subjects separately. This will be performed based on the total number of firings. An intervention is defined as any firing which is classified as hemostasis intervention. To establish that the intervention rate is not increased compared to SOC, a 95% confidence interval for the difference in proportion of firings requiring interventions for PVS minus SOC will be calculated and powered vascular stapler will be considered to have acceptable performance if the upper bound of the 95% confidence interval does not exceed 3%.

Additional endpoints will be summarized with descriptive statistics and 95% confidence intervals as appropriate for continuous or categorical measurements.

#### 7.5 STATISTICAL/ANALYTICAL ISSUES

#### 7.5.1 Handling of Dropouts or Missing Data

All summaries will be performed only on subjects undergoing the surgical procedure and only observed data will be summarized. There will be no imputation of data for early terminated subjects or for missing data within the database.

# 7.5.2 Interim Analyses and Data Monitoring

No interim analysis is planned for this study.

#### 7.5.3 Multicenter Studies

No adjustment for center is planned in the statistical analysis. Center specific analyses may be conducted pending within-center sample size to understand the effect that surgeon techniques and site standard of care may have on the overall results.

## 7.5.4 Multiple Comparisons/Multiplicity

No adjustment for multiplicity is necessary since multiple hypotheses are not being tested.

#### 7.6 ANALYSIS OF SAFETY

The number and percentage of subjects requiring hemostasis interventions postoperatively that are classified as related to SOC/PVS for RA/RV transection (e.g. need for blood product transfusion or additional surgical procedure) will be summarized for each

Protocol ESC-15-002 Version/Date: Original/17 NOV2015 FINAL



group as a primary safety endpoint.

Safety will be assessed through the incidence of AEs and serious adverse events (SAEs), which will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs will be summarized at the MedDRA system organ class and preferred term level. Incidence of AEs will also be summarized by maximum severity. All reported adverse events will be listed.

# 8.0 RISKS AND BENEFITS OF THE STUDY DEVICE AND CLINICAL INVESTIGATION

The procedure being performed with powered vascular stapler is identical to the procedure subjects would receive as part of their standard of care procedure. To date, no risks have been reported beyond standard risks associated with simple laparoscopic nephrectomies and laparoscopic nephroureterectomies. This study may or may not provide any benefits to the subject.

### 9.0 ADVERSE EVENTS AND PRODUCT COMPLAINTS

#### 9.1 DEFINITIONS

#### 9.1.1 Adverse Event

An adverse event is defined as any undesirable clinical occurrence in a subject that may or may not be attributable to the device or procedure. All AEs, regardless of their relationship to the procedure or device, are to be recorded in the eCRF and reported to the Sponsor.

In addition, the Investigator is required to provide:

- The onset and resolution dates of the event;
- The severity of the event;
- The outcome of the event:
- The relationship of the event to procedure and/or device (ECHELON FLEX™ Powered Vascular Stapler with Advanced Placement Tip or standard of care stapler); and
- The action taken for the medical management of the event.

Postoperative pain is expected and will not be documented as an adverse event unless the Investigator considers the pain to exceed what is typically anticipated following a laparoscopic nephrectomy or laparoscopic nephroureterectomy. (This data is separate from incisional and/or trocar pain).

# 9.1.2 Anticipated Adverse Events

An expected morbidity/procedural complication is defined as an AE that is known to be common or usual in nature, severity, or incidence during laparoscopic nephrectomies/ nephroureterectomies.

A list of anticipated AEs that may occur during this study are listed in Appendix I.

### 9.1.3 Serious Adverse Event

It is the Investigator's responsibility to determine if an AE is an SAE.

Protocol ESC-15-002 

Version/Date: Original/17 NOV2015 FINAL



#### SAEs are AEs that:

- Led to death,
- Led to serious deterioration in the health of the subject, that either resulted in
  - a life-threatening illness or injury, or
  - a permanent impairment of a body structure or a body function, or
  - in-patient or prolonged hospitalization, or
  - medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  - Led to fetal distress, fetal death or a congenital abnormality or birth defect

Note: "Death" should not be reported as an adverse event. The cause of death should be reported as an adverse event. The only exception is "Sudden Death" when the cause is unknown.

# 9.1.4 Severity of Adverse Events

It is the Investigator's responsibility to assess the severity of an AE. A change in severity may constitute a new reportable AE.

The following guideline should be used to determine the severity of each adverse event:

- MILD: Awareness of experience, but easily tolerated. No medical intervention required.
- MODERATE: Enough discomfort to interfere with usual activities. Medical intervention required.
- **SEVERE**: Inability to carry out usual activities. Medical intervention (including hospitalization or prolongation of hospitalization) required.

### 9.1.5 Relationship of Adverse Events

It is the Investigator's responsibility to assess the relationship of an AE to the study procedure (laparoscopic nephrectomies/ nephroureterectomies) and powered vascular stapler or SOC.

The following guidelines should be used in determining the relationship of an adverse event to the study device, study procedure, or other causality:

- Not Related A clinical event (including abnormal laboratory result) that results from causes extraneous to administration of device/procedure/other and is most likely due to alternative etiology, (i.e., pre-existing condition, underlying disease, intercurrent illness, concomitant medications);
- Possibly A clinical event (including abnormal laboratory result) that presents an unlikely association between device/procedure/other, which cannot be ruled out with certainty, but could also be explained by alternative etiology;
- Related

   A clinical event (including abnormal laboratory result) that presents a



- strong temporal relationship between device/procedure/other, in which an alternative etiology is unlikely; or
- Unknown A clinical event (including abnormal laboratory result) that cannot be determined to be related or unrelated to device/procedure/other given the information obtained.

# 9.1.6 Product Complaints

A product complaint is defined as any written, electronic or oral communication that alleges deficiencies related to the identity, labeling, quality, durability, reliability, safety, effectiveness, or performance of a device (i.e., stapler) after it is released for distribution (policy of Johnson and Johnson Medical Device Quality management). A product complaint may or may not be associated with an AE/SAE.

# 9.2 REPORTING PROCEDURES FOR ADVERSE EVENTS/PRODUCT COMPLAINTS

# 9.2.1 Reporting Adverse Events

Data related to AEs will be recorded in the source documentation from the time of study enrollment (first incision) until the subject completes the study or terminates early. All AEs that are unresolved at study completion (or early termination) will be recorded as ongoing at study end.

Data related to SAEs will be collected until event resolution, or until the event is considered stable, or until all attempts to determine the resolution of the event are exhausted.

# 9.2.2 Reporting Serious Adverse Events

The site must complete the SAE eCRF within 24 hours of becoming aware of the event.

Supporting SAE documentation can be faxed to:



The Investigator will also be required to assess if the SAE is considered anticipated (see Appendix I) and if the event involved a product complaint. The report of an SAE by a study site does not constitute an admission that study personnel or the user facility (hospital/clinic) caused or contributed to the event.

The study site is also responsible for submitting to the reviewing IRB/EC according to their IRB/EC procedures.

Protocol ESC-15-002 

Version/Date: Original/17 NOV2015 FINAL



# 9.2.3 Reporting Product Complaints

All product complaints related to powered vascular stapler shall be documented throughout the clinical investigation.

Product complaints related to powered vascular stapler must be reported to the Sponsor in a timely manner and no later than 24 hours after becoming aware of the event. The Product Complaint Form must be emailed to the EES Customer Complaint team at the following email address:

One copy of the processed form should be kept on-site and the device should be retained. EES representatives will organize collection of the device for evaluation as needed.

#### 10.0 REFERENCE LIST

- 1. Santucci, R., Al-Qudah, H., (2013) "Radical Nephrectomy", Medscape, accessed March 5, 2015, http://emedicine.medscape.com/article/448878-overview#showall
- "Cancer Facts & Figures 2014", American Cancer Society, Inc., accessed March 5, 2015, <a href="http://www.cancer.org/acs/groups/content/%40research/documents/webcontent/acspc-042151.pdf">http://www.cancer.org/acs/groups/content/%40research/documents/webcontent/acspc-042151.pdf</a>
- 3. Su, L., Ratner, L., Montgomery, R., Jarrett, T., Trock, B., Sinkov, V., Bluebond-Langner, R., Kavoussi, L (2004, Aug). Annals of Surgery, Volume 240(2): 358-363
- 4. Burgess, N. A., Koo, B. C, Calvert, R. C., Hindmarsh, A, Donaldson, P.J., Rhodes, M. (2007). Journal of Endourology; Volume 21, Issue 6: 610-613

Protocol ESC-15-002 



# **APPENDIX I: ANTICIPATED ADVERSE EVENTS**

| Associated with Surgery and<br>General Anesthesia | Simple/Radical Laparoscopic Nephrectomy or<br>Laparoscopic Nephroureterectomy Surgery<br>Specific |
|---|---|
| Acute Lung Injury | Air/Gas Embolism |
| Acute Respiratory Distress Syndrome | Chylothorax |
| Adhesions | Diaphragmatic Injury |
| Altered Mental Status | Emphysema |
| Anaphylaxis | Esophageal Injury |
| Anemia | Incisional hernia |
| Angina | Injury to other organs |
| Atelectasis | Intercostal nerve injury |
| Bacteremia | Internal Hernia |
| Bleeding | Pneumothorax |
| Bradycardia | Small bowel obstruction |
| Cardiac Arrhythmia | Splenic injury |
| Central line infection | Thromboembolic Event |
| Cerebrovascular Accident / Stroke | Wound infection |
| Congestive Heart Failure | |
| Constipation | |
| Death | |
| Deep Venous Thrombosis | |
| Dehydration | |
| Dementia | |
| Diarrhea | |
| DIC, Coagulopathy | |
| Dizziness | |
| Dyspnea | |
| Electrolyte Imbalance | |
| Fever, Pyrexia | |
| Headache | |
| Hematoma | |
| Hematuria | |
| Hypertension | |
| Hypotension, shock | |
| Нурохіа | |
| lleus | |
| Infection/SSI/Abscess | |
| Jaundice | |
| Lethargy | |
| Leukocytosis | |

Protocol ESC-15-002 Version/Date: Original/17 NOV2015 FINAL



| Liver Failure |
|-----------------------------------------------|
| Mesenteric Infarct |
| Mesenteric Ischemia |
| Myocardial Infarction |
| Nausea |
| Obtundation, Depressed Level of Consciousness |
| Oliguria |
| Pain (increased/severe/chronic) |
| Pneumonia |
| Port Site Hernia |
| Pulmonary Edema |
| Pulmonary Embolism |
| Renal Failure |
| Respiratory Failure |
| Respiratory Insufficiency |
| Sepsis |
| Somnolence |
| Systemic Inflammatory Response Syndrome |
| Tachycardia |
| Thrombocytopenia |
| Thromboembolic Event |
| Thrombosis |
| TIA |
| Tightness of the chest, Angina |
| Tinnitus |
| Urinary Retention |
| Urinary Tract Infection (UTI) |
| Volume Depletion, Hypovolemia |
| Vomiting |
| Wheezing |
| Wound Dehiscence |